CLINICAL TRIAL: NCT01655927
Title: PHASE 3 STUDY OF EFFICACY OF TRANEXAMIC ACID IN BRAIN TUMORS RESECTIONS
Brief Title: Efficacy of Tranexamic Acid in Brain Tumor Resections
Acronym: COLFIRE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colombian Foundation for Epilepsy and Neurological Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT28072012FIRE
Record Dates: First submitted 2012-07-30; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Brain Tumors; Neoplasms; Gliomas; Astrocytomas; Meningiomas
Keywords: Neoplasms; Tranexamic Acid; Brain Tumors
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Glioma; Astrocytoma; Meningioma | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): 15 mg/Kg Tranexamic Acid IV after anesthesic induction,and continues with a dose of 1mg/kg/h intraoperatory
  Interventions: Drug: Tranexamic Acid
- Saline (Placebo) (Placebo Comparator): 15 mg/Kg of Saline IV after anesthesic induction,and continues with a dose of 1mg/kg/h intraoperatory
  Interventions: Drug: Placebo: Saline

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Drug: Placebo: Saline
  Arms: Saline (Placebo)

SUMMARY:
The purpose of this study is to determine whether Tranexamic Acid is effective or not in the reduction of intraoperative bleeding loss in brain tumors resections.

DETAILED DESCRIPTION:
Brain tumor resection has been associated with increased blood loss and a significant increase in the incidence of Intravascular disseminated coagulopathy. The development of coagulopathy in the context of tumor resection is associated with poor results. Transfusion decision during the course of neurosurgical surgery offers benefits such as increased oxygen carrying capacity but may increase the risk associated with transfusions such as blood infections, hemolysis, lung injury and immunosuppression. The information available on tranexamic acid used in neurosurgery is little, therefore this opens up new alternatives in the techniques of reducing intraoperative bleeding.

Tranexamic acid is an antifibrinolytic agent that blocks the binding of plasminogen to the fibrin surface. It has been used to reduce blood loss during coronary revascularization, liver resection, obstetrics and orthopedic procedures. Tranexamic acid intraoperatively has been shown to reduce blood loss up to 45%. The primary concern when administering an antifibrinolytic drug is the potential increased incidence of thromboembolic events. There is no actual data on the utility of tranexamic acid to reduce blood loss in brain tumors resection surgery.

We want to compare Tranexamic Acid to Saline solution(Placebo) to see whether Tranexamic ACid Administration will reduce blood loss during brain tumor resection. Reduction in transfusion requirements will lead to reduced costs and possible reduction in complications of blood transfusion and perioperative incidents.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate by giving informed consent
* Eligible previously untreated patients with resectable brain tumor.

Exclusion Criteria:

* Patients with previous thromboembolic events.
* Patients with coagulopathy or anticoagulation therapy. (Abnormal PT, PTT)
* Patients with impaired renal function (Creatinine >1.1mg/dl)
* Patients with known contraindications to fibrinolytic treatment.
* Patients receiving rejection therapy.
* Patients with abnormal liver function.
* Known allergies to Tranexamic Acid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with need of blood transfusion. | 24-48 hours
  (Measured with Hemoglobin/Hematocrit, PT, PTT, Plackets: pre-surgery, 6 hrs after surgery and 24 hours after.)

CONTACTS AND LOCATIONS:
Overall Officials: Randy O Guerra, MD, Study Director — Colombian foundation center for epilepsy and neurological disease - FIRE; Fredy Diaz, MD, Principal Investigator — Colombian foundation center for epilepsy and neurological disease -FIRE
Locations (1):
- Colombian foundation center for epilepsy and neurological disease, Cartagena, Departamento de Bolívar, Colombia